CLINICAL TRIAL: NCT05831137
Title: The Optimization of the Intercostal Nerves Cryoablation Aplication Time During Nuss Procedure
Brief Title: Cryoanalgesia Aplication Time Optimization During Nuss Procedure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PUM NUSS
Record Dates: First submitted 2023-04-04; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-03

CONDITIONS: Funnel Chest; Excavatum, Pectus
Keywords: nuss procedure; cryoanalgesia
MeSH Terms: conditions — Funnel Chest

STUDY DESIGN:
Intervention Model Description: In each patient one side of the chest will be treated by standard metod and the second side will be treated with the novel method.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention side (Experimental): duration of intercostal nerves cryolesia: 1 minute per left nerve
  Interventions: Procedure: shorter cryoanalgesia
- control side (No Intervention): duration of intercostal nerves cryolesia: 2 minute per right nerve

INTERVENTIONS:
Procedure: shorter cryoanalgesia — duration time of cryoanalgesia
  Arms: intervention side

SUMMARY:
This study compared standard therapy (multimodal analgesia with 2 minutes cryoanalgesia) versus a novel approach (multimodal analgesia with 1 minute cryoanalgesia) in subject undergoing minimal invasive modyfied Nuss procedure with thoracoscopy.

DETAILED DESCRIPTION:
Funnel chest deformation may be a great challenge for therapeutic teams due to severe pain in the postoperative period as well as chronic pain.

2 minutes per one intercostal nerve aplication cryoanalgesia as a part of multimodal analgesia is a standard protocol in many countries.

This Prospective Non-Randomized Study is a single institution pilot study designed to compare standard therapy (control side: multimodal analgesia with 2 minutes cryoanalgesia) versus a novel approach (multimodal analgesia with 1 minute cryoanalgesia) in each patient to address the need for better management of acute and long-term pain in the pediatric population diagnosed with funnel-chest and treated using the modyfied Nuss method.

All of the patients will receive a standard care according to Polish guidelines: multimodal analgesia with regional analgesia (bilateral erector spine plane block) with cryoanalgesia. The right intercostal nerves will be treated with 2 minutes cryoanalgesia (control side). The left side of the chest (left intercostal nerves) will be treated with 1 minute cryoanalgesia (intervention side).

The intraoperative cryoanalgesia will be performed using the Cryo-S Painless device (Metrum - Cryoflex Polska Limited).

The study will assess the effectiveness of shorter aplication duration time of cryoanalgesia as a method of acute and long-term pain control and safety of the method.

Specific Aim: To determine if, compared with current 2 minutes cryoanalgesia protocol, 1 minute aplication time of cryoanalgesia is effective at the same level when consider pain control and postoperative functioning in each patient.

The results were compared in terms of demographics, right versus left side of the chest pain levels, quality and length of rehabilitation and patient satisfaction using the Quality of Life by modyfied Nuss questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing pectus excavatum repair with modyfied minimal invasive thoracoscopic Nuss technique
* informed concent signed for cryolesia

Exclusion Criteria:

* age 9 years or below
* refuse to receive cryoanalgesia or regional anaesthesia as a primary pain relief

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2023-06-10 (Estimated); Study Completion 2023-07-10 (Estimated)

PRIMARY OUTCOMES:
The worse pain occurrence during first 24 hours after operation. | up to 24 hours after operation
  numeric pain score, range from 0 to 10

SECONDARY OUTCOMES:
thoracic hypoaesthesia occurrence | up to 24 hours after operation
  cold test assessment (yes / no)
residual wound or chest pain occurrence | postoperative months 1,3
  the chest or wound chronic pain occurrence
duration of hospitalization | estimated 4 days
  the lengh of the time in days spent in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Jowita Biernawska, MD PhD, Study Director — Pomeranian Medical Universitet Szczecin
Locations (1):
- Pomeranian Medical University, Szczecin, Poland

IPD SHARING:
Plan to Share IPD: Yes
We invite others researchers to collaboration as multicenter study
Supporting Information: Study Protocol
Time Frame: up to 12 months from the beginning of the study
Access Criteria: by contacy to the Principal Investigator

REFERENCES:
- [Result] Zeineddin S, Goldstein SD, Linton S, DeBoer C, Alayleh A, Ortiz I, Sands L, Kujawa S, Suresh S, Ghomrawi H, Abdullah F. Effectiveness of one minute per level intercostal nerve cryoablation for postoperative analgesia after surgical correction of pectus excavatum. J Pediatr Surg. 2023 Jan;58(1):34-40. doi: 10.1016/j.jpedsurg.2022.09.032. Epub 2022 Sep 26. PMID 36283847